CLINICAL TRIAL: NCT04928846
Title: A Phase 3 Open-Label, Randomized, Controlled, Global Study of Telisotuzumab Vedotin (ABBV-399) Versus Docetaxel in Subjects With Previously Treated c-Met Overexpressing, EGFR Wildtype, Locally Advanced/Metastatic Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study to Assess Disease Activity and Adverse Events of Intravenous (IV) Telisotuzumab Vedotin Compared to IV Docetaxel in Adult Participants With Previously Treated Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M18-868; 2023-505749-14-00 (Other: EU CT)
Expanded Access: NCT04830202 (Available)
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: c-Met Overexpressing Non-Small Cell Lung Cancer; c-Met NSCLC; Telisotuzumab Vedotin; ABBV-399; Docetaxel; Cancer; Non Small Cell Lung Cancer; NSCLC; TeliMET NSCLC-01; Teliso-V
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — telisotuzumab vedotin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Telisotuzumab Vedotin (Experimental): Participants will receive telisotuzumab vedotin every 2 weeks until meeting study drug discontinuation criteria.
  Interventions: Biological: Telisotuzumab Vedotin
- Docetaxel (Active Comparator): Participants will receive docetaxel every 3 weeks until meeting study drug discontinuation criteria.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Telisotuzumab Vedotin — Intravenous (IV) Infusion
  Other Names: ABBV-399
  Arms: Telisotuzumab Vedotin
Drug: Docetaxel — IV Infusion
  Arms: Docetaxel

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. Non-small cell lung cancer (NSCLC) is a solid tumor, a disease in which cancer cells form in the tissues of the lung. The purpose of this study is to determine if telisotuzumab vedotin works better than docetaxel and to assess how safe telisotuzumab vedotin is in adult participants with NSCLC who have previously been treated. Change in disease activity and adverse events will be assessed.

Telisotuzumab vedotin is an investigational drug being developed for the treatment of NSCLC. Participants will be randomly assigned a treatment of Teliso-V or Docetax at an 1:1 ratio. Each group receives intravenous (IV) infusion of telisotuzumab vedotin or IV infusion of docetaxel. Approximately 698 adult participants with c-Met overexpressing NSCLC will be enrolled in the study in approximately 330 sites worldwide.

Participants will receive IV telisotuzumab vedotin every 2 weeks or docetaxel every 3 weeks until meeting study drug discontinuation criteria. At the conclusion of the study, participants who continue to demonstrate clinical benefit may be eligible to receive study treatment via an extension of the study, a rollover study, or through another mechanism.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Projected life expectancy of at least 12 weeks.
* Participants must have c-Met overexpressing non-small cell lung cancer (NSCLC) as assessed by an AbbVie designated immunohistochemistry (IHC) laboratory using the VENTANA MET (SP44) RxDx assay.
* Archival or fresh tumor material must be submitted for assessment of c-Met protein expression levels during the Pre-Screening period. Tumor material from the primary tumor site and/or metastatic sites are allowed.

  * If a participant was prescreened for Study M14-239 but did not enroll, tumor material previously submitted for Study M14-239 may be used for Study M18-868 Pre-Screening upon confirmation from AbbVie that sufficient evaluable tumor material is available (Except China).
* A histologically or cytologically documented non-squamous cell NSCLC that is locally advanced or metastatic.
* A known epidermal growth factor receptor (EGFR) activating mutation status.

  -- Participants with actionable EGFR activating mutations are not eligible
* Actionable alterations in genes other than EGFR are eligible.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Have received no more than 1 line of prior systemic cytotoxic chemotherapy in the locally advanced or metastatic setting.

  * Neoadjuvant and adjuvant systemic cytotoxic chemotherapy will count as a prior line for eligibility purposes if progression occurred within 6 months of the end of therapy.
* Have progressed on at least 1 line of prior therapy for locally advanced/metastatic NSCLC:

  * Participants WITHOUT an actionable gene alteration: must have progressed on (or be considered ineligible for) platinum-based chemotherapy and immune checkpoint inhibitor (as monotherapy or in combination with chemotherapy).
  * Participants WITH an actionable gene alteration for which immune checkpoint inhibitor therapy is not standard of care (e.g., anaplastic lymphoma kinase [ALK] translocation): must have progressed on (or be considered ineligible for) anti-cancer therapy targeting driver gene alterations and platinum-based chemotherapy.

    * Participants with actionable gene alterations for which immune checkpoint inhibitor is standard of care must have also progressed on (or be considered ineligible for) immune checkpoint inhibitor (as monotherapy or in combination with chemotherapy).
* Must be considered appropriate for docetaxel therapy based on the assessment of the treating physician.
* Participants with metastases to the central nervous system (CNS) are eligible only after adequate treatment (such as surgery, radiotherapy, or drug therapy) is provided and:

  * They are asymptomatic and off or on a stable or reducing dose of systemic steroids (on no more than 10 mg per day [QD] prednisone or equivalent) and/or anticonvulsants for at least 2 weeks prior to randomization.

Exclusion Criteria:

* Evidence of new, untreated CNS metastases or progressing CNS metastases after treatment.
* Evidence of leptomeningeal disease.
* Participants with adenosquamous or neuroendocrine histology, nor sarcomatoid features.
* Epidermal growth factor receptor (EGFR) activating mutations.
* Participants who have received prior c-Met-targeted antibodies, prior telisotuzumab vedotin, or prior antibody-drug conjugates either targeting c-Met or consisting of monomethylauristatin E..
* Participants who have received prior docetaxel therapy.
* A history of other malignancies except:

  * Malignancy treated with curative intent and with no known active disease present for >=2 years before the first dose of study drug and felt to be at low risk for recurrence by investigator. Additionally, participants must not be receiving any ongoing anti-cancer therapy, including maintenance therapy, prior to randomization..
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without current evidence of disease.
* A history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. A history of prior radiation pneumonitis in the radiation field (fibrosis) is not permitted.
* Unresolved or neuroendocrine histology, nor sarcomatoid features adverse event (AE) >= Grade 2 from prior anticancer therapy, except for alopecia or anemia. Participants with hormone deficiencies caused by prior anticancer therapy who are asymptomatic and on a stable dose of replacement hormone are eligible for study.
* Major surgery within 21 days prior to randomization.
* Clinically significant condition(s) as listed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) per Blinded Independent Central Review (BICR) | Up to approximately 39 months
  PFS is defined as the time from randomization to the first occurrence of radiographic progression based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) per BICR or death from any cause.
Overall Survival (OS) | Up to approximately 39 months
  OS is defined as the time from randomization to the event of death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR), per BICR. | Up to approximately 58.25 months
  ORR is defined as the proportion of participants with a complete response (CR) or partial response (PR) based on RECIST v1.1
Duration of Response (DoR), per BICR | Up to approximately 58.25 months
  DoR is defined for responders as the time from response (CR or PR) to the first occurrence of radiographic progression per RECIST v1.1 or death from any cause.
PFS per Investigator Assessment | Up to approximately 58.25 months
  PFS is defined as the time from randomization to the first occurrence of radiographic progression based on RECIST version 1.1 per investigator or death from any cause. Participants with no PFS event will be censored at the last evaluable radiographic assessment per investigator. Participants with no event and no evaluable post-baseline assessment will be censored at randomization.
Change from Baseline of Physical Functioning as measured by the Physical Functioning domain of the EORTC-QLQ-Core 30 (EORTC QLQ-C30). | Up to approximately 12 Weeks
  The EORTC QLQ-C30 assesses health-related quality of life in cancer patients participating in clinical trials. The EORTC QLQ-C30 comprises 5 functional scales (physical, role, emotional, social, cognitive), 8 single-item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, and dyspnea), as well as subscales assessing global health/quality of life and financial impact. Raw scores are transformed to a scale of 0 to 100, with higher scores representing better functioning/quality of life and greater symptom burden.
Change from Baseline in Quality of Life as measured by the Global Health Status/Quality of Life Domain of the EORTC QLQ-C30. | Up to approximately 12 Weeks
  The EORTC QLQ-C30 assesses health-related quality of life in cancer patients participating in clinical trials. The EORTC QLQ-C30 comprises 5 functional scales (physical, role, emotional, social, cognitive), 8 single-item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, and dyspnea), as well as subscales assessing global health/quality of life and financial impact. Raw scores are transformed to a scale of 0 to 100, with higher scores representing better functioning/quality of life and greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (314):
- United States (50):
  - University of Alabama at Birmingham - Main /ID# 247074, Birmingham, Alabama
  - Ironwood Cancer & Res Ctr /ID# 262446, Chandler, Arizona
  - Mayo Clinic Arizona /ID# 255858, Phoenix, Arizona
  - Onvida Health Yuma Medical Center /ID# 253625, Yuma, Arizona
  - City of Hope /ID# 243157, Duarte, California
  - City Of Hope - Seacliff /ID# 263143, Huntington Beach, California
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 263144, Irvine, California
  - City Of Hope - Antelope Valley /ID# 263138, Lancaster, California
  - The Oncology Institute Of Hope & Innovation -East Los A /ID# 239774, Los Angeles, California
  - University of California, Los Angeles /ID# 253954, Los Angeles, California
  - Eisenhower Medical Center /ID# 233189, Rancho Mirage, California
  - Mayo Clinic Hospital Jacksonville /ID# 254688, Jacksonville, Florida
  - Ocala Oncology Florida Cancer Affiliates - Main /ID# 234228, Ocala, Florida
  - BRCR Medical Center Inc /ID# 262344, Tamarac, Florida
  - Memorial University Medical Center /ID# 264081, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center /ID# 238363, Honolulu, Hawaii
  - Edward-Elmhurst Cancer Center /ID# 238552, Elmhurst, Illinois
  - Springfield Clinic - First /ID# 262290, Springfield, Illinois
  - Goshen Center for Cancer Care /ID# 257734, Goshen, Indiana
  - Investigative Clinical Research of Indiana - Indianapolis /ID# 260468, Indianapolis, Indiana
  - Baptist Health Lexington /ID# 252769, Lexington, Kentucky
  - Dana-Farber Cancer Institute /ID# 247132, Boston, Massachusetts
  - Trinity Health St. Joseph Mercy Ann Arbor /ID# 232190, Ypsilanti, Michigan
  - Mayo Clinic - Rochester /ID# 252052, Rochester, Minnesota
  - Hattiesburg Clinic /ID# 248033, Hattiesburg, Mississippi
  - St. Luke's Hospital - Chesterfield /ID# 251688, Chesterfield, Missouri
  - St. Lukes Hosp. of Kansas City /ID# 259940, Kansas City, Missouri
  - Alliance for Multispecialty Research (AMR) - Kansas City /ID# 247567, Kansas City, Missouri
  - Hulston Cancer Center /ID# 232226, Springfield, Missouri
  - Saint Louis University Cancer Center /ID# 260722, St Louis, Missouri
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana /ID# 253147, Billings, Montana
  - Nebraska Hematology Oncology /ID# 257710, Lincoln, Nebraska
  - Renown Medical Group - Oncology/Hematology /ID# 247942, Reno, Nevada
  - Astera Cancer Care /ID# 257753, East Brunswick, New Jersey
  - San Juan Oncology Associates /ID# 244387, Farmington, New Mexico
  - Maimonides Medical Center /ID# 240783, Brooklyn, New York
  - Northwell Health - Monter Cancer Center /ID# 247081, Lake Success, New York
  - AdventHealth Hendersonville /ID# 265349, Hendersonville, North Carolina
  - FirstHealth of the Carolinas- Speciality Center /ID# 241279, Pinehurst, North Carolina
  - Genesis Cancer Care Center /ID# 239190, Zanesville, Ohio
  - Cancer Care Associates Of York /ID# 266143, York, Pennsylvania
  - Medical University of South Carolina /ID# 251383, Charleston, South Carolina
  - St Francis Cancer Center /ID# 243596, Greenville, South Carolina
  - Avera Cancer Institute - Aberdeen /ID# 257759, Aberdeen, South Dakota
  - Avera Cancer Institute /ID# 239635, Sioux Falls, South Dakota
  - Duplicate_Memphis VA Medical Center /ID# 263250, Memphis, Tennessee
  - Dell Seton Medical Center /ID# 247016, Austin, Texas
  - Community Cancer Trials of Utah - South Ogden /ID# 262829, Ogden, Utah
  - Valley Medical Center /ID# 253950, Renton, Washington
  - Medical Oncology Associates /ID# 247003, Spokane, Washington
- Argentina (6):
  - Cemic /Id# 231486, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires /ID# 231495, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Centro Médico Austral /ID# 239860, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Clinicas Clinica Viedma S.A. /ID# 232339, Viedma, Río Negro Province
  - LC Investigacion /ID# 239880, Buenos Aires
  - Instituto de Oncología Angel H. Roffo /ID# 231499, Buenos Aires
- Australia (4):
  - Port Macquarie Base Hospital /ID# 273654, Port Macquarie, New South Wales
  - Westmead Hospital /ID# 274447, Westmead, New South Wales
  - Barwon Health /ID# 241920, Geelong, Victoria
  - Austin Health /ID# 247507, Heidelberg, Victoria
- Austria (8):
  - Medizinische Universitaet Innsbruck /ID# 240981, Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 240967, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH /ID# 249000, Wels, Upper Austria
  - Medizinische Universitaet Wien /ID# 230615, Vienna, Vienna
  - Klinik Penzing /ID# 230700, Vienna, Vienna
  - Klinik Floridsdorf /ID# 230608, Vienna, Vienna
  - Landeskrankenhaus Feldkirch /ID# 250333, Feldkirch, Vorarlberg
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 232467, Salzburg
- Belgium (10):
  - Algemeen Ziekenhuis klina /ID# 239853, Brasschaat, Antwerpen
  - Universitair Ziekenhuis Antwerpen /ID# 239971, Edegem, Antwerpen
  - Grand Hôpital de Charleroi - Les Viviers /ID# 234178, Charleroi, Hainaut
  - Hospital La Louviere Site Jolimont - Helora /ID# 246771, La Louvière, Hainaut
  - Jessa Ziekenhuis /ID# 246766, Hasselt, Limburg
  - Vitaz /Id# 246773, Sint-Niklaas, Oost-Vlaanderen
  - Institut Jules Bordet /ID# 246770, Anderlecht
  - AZ Maria Middelares /ID# 246768, Ghent
  - CHU de Liege /ID# 246772, Liège
  - UCL Namur University Hospital, Site Sainte-Elisabeth /ID# 246769, Namur
- Brazil (9):
  - Ensino e Terapia de Inovacao - Clinica AMO /ID# 231604, Salvador, Estado de Bahia
  - Irmandade da Santa Casa de Misericordia de Porto Alegre /ID# 233249, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos /ID# 233247, Barretos, São Paulo
  - OC Oncoclínicas SP /ID# 261828, São Paulo, São Paulo
  - Instituto Nacional de Cancer (INCA) /ID# 231509, Rio de Janeiro
  - Instituto Dor de Pesquisa e Ensino /ID# 233245, Rio de Janeiro
  - Instituto de Ensino e Pesquisas Sao Lucas /ID# 247417, São Paulo
  - Hospital Sirio Libanes /ID# 261827, São Paulo
  - Casa de Saúde Santa Marcelina /ID# 231605, São Paulo
- Bulgaria (5):
  - Mbal Uni Hospital /ID# 273707, Panagyurishte, Pazardzhik
  - University Multiprofile Hospital for Active Treatment Sofiamed /ID# 234108, Sofiya, Sofia
  - Complex Oncology Center - Burgas /ID# 240532, Burgas
  - Complex Cancer Center Plovdiv /ID# 234106, Plovdiv
  - UMHAT Multiprofile Hospital for Active Treatment Sveta Marina /ID# 234112, Varna
- Canada (5):
  - Cross Cancer Institute /ID# 252065, Edmonton, Alberta
  - William Osler Health System - Brampton Civic Hospital /ID# 254420, Brampton, Ontario
  - CISSS de la Monteregie /ID# 239081, Greenfield Park, Quebec
  - CSSS Alphonse-Desjardins, CHAU de Levis /ID# 261158, Lévis, Quebec
  - Hopital Du Sacre-Coeur De Montreal /ID# 274584, Montreal, Quebec
- Chile (6):
  - Clinica Universidad Catolica del Maule /ID# 231294, Talca, Maule Region
  - Icegclinic /Id# 231212, La Florida, Santiago Metropolitan
  - Sociedad Prosalud Montes y Orlandi /ID# 231154, Providencia, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez /ID# 231151, Providencia, Santiago Metropolitan
  - Sociedad Oncovida /ID# 231152, Providencia, Santiago Metropolitan
  - Hospital Clinico Universidad De Los Andes /ID# 260974, Santiago
- China (45):
  - Anhui Medical University - Anhui Chest Hospital /ID# 231899, Hefei, Anhui
  - Beijing Cancer Hospital /ID# 231923, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital (East) - Dongdan Campus /ID# 233175, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University /ID# 232202, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University /ID# 251592, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital /ID# 243134, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University /ID# 242381, Xiamen, Fujian
  - The First Affiliated Hospital Of Guangzhou Medical University /ID# 238591, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College /ID# 242182, Shantou, Guangdong
  - Affiliated Hospital of Guangdong Medical College /ID# 233317, Zhanjiang, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University /ID# 231855, Nanning, Guangxi
  - People's Hospital of Guizhou Province /ID# 243614, Guiyang, Guizhou
  - Affiliated Hospital of Hebei University /ID# 239586, Baoding, Hebei
  - Harbin Medical University Cancer Hospital /Id# 231941, Harbin, Heilongjiang
  - The First affiliated Hospital of Nanyang Medical College /ID# 244652, Nanyang, Henan
  - People's Hospital of Henan Province /ID# 242187, Zhengzhou, Henan
  - Henan Cancer Hospital /ID# 239577, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 231904, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST /ID# 239575, Wuhan, Hubei
  - Hubei Cancer Hospital /ID# 240045, Wuhan, Hubei
  - Hunan Cancer Hospital /ID# 231943, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University /ID# 242179, Hohhot, Inner Mongolia
  - Nanjing Drum Tower Hospital /ID# 231791, Nanjing, Jiangsu
  - Nantong Tumor Hospital /ID# 232424, Nantong, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 231934, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University /ID# 231935, Nanchang, Jiangxi
  - Jilin Cancer Hospital /ID# 244702, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University /ID# 239755, Dalian, Liaoning
  - First Affiliated Hospital of China Medical University /ID# 231924, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University /ID# 232023, Xi'an, Shaanxi
  - Shandong University - Jinan Central Hospital /ID# 231895, Jinan, Shandong
  - Shandong Cancer Hospital /ID# 251506, Jinan, Shandong
  - LinYi Cancer Hospital /ID# 239713, Linyi, Shandong
  - Shanghai Chest Hospital /ID# 231897, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital /ID# 258674, Taiyuan, Shanxi
  - Sichuan Cancer Hospital /ID# 239707, Chengdu, Sichuan
  - West China Hospital, Sichuan University /ID# 233703, Chengdu, Sichuan
  - Tianjin Cancer Hospital /ID# 233176, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital /ID# 231839, Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital of Xinjiang Medical University /ID# 240094, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital /ID# 251388, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 232032, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital /ID# 242476, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province /ID# 232021, Linhai, Zhejiang
  - Ningbo No. 2 Hospital /ID# 242478, Ningbo, Zhejiang
- Colombia (4):
  - Hospital Pablo Tobón Uribe /ID# 258128, Medellín, Antioquia
  - Fundación Ctic - Centro De Tratamiento E Investigación Sobre Cáncer Luis Carlos /ID# 258131, Bogotá, Bogota D.C.
  - Sociedad de Oncologia y Hematologia del Cesar SAS /ID# 258130, Valledupar, Cesar Department
  - Imat Oncomedica /ID# 258129, Montería, Departamento de Córdoba
- Czechia (2):
  - Masarykuv onkologicky ustav /ID# 232426, Brno
  - Nemocnice AGEL Novy Jicin, a.s. /ID# 232427, Nový Jičín
- Denmark (2):
  - Roskilde Sygehus /ID# 241842, Roskilde, Region Sjælland
  - Odense University Hospital /ID# 241663, Odense, Region Syddanmark
- France (12):
  - APHM - Hopital Nord /ID# 251935, Marseille, Bouches-du-Rhone
  - CHU Lille - Hôpital Albert Calmette /ID# 251934, Lille, Hauts-de-France
  - Hopital Arnaud de Villeneuve /ID# 239404, Montpellier, Herault
  - Centre Hospitalier Universitaire de Bordeaux /ID# 244953, Pessac, Nouvelle-Aquitaine
  - Institut Curie /ID# 240141, Paris, Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin /ID# 239409, Paris, Paris
  - Centre Hospitalier d'Avignon /ID# 275229, Avignon, Provence-Alpes-Côte d'Azur Region
  - Hospices Civils de Lyon (HCL) - Hopital Louis Pradel /ID# 251933, Bron, Rhone
  - Centre Leon Berard /ID# 267397, Lyon, Rhone
  - Centre Hosp Intercommunal de Creteil /ID# 251936, Créteil, Val-de-Marne
  - AP-HP - Hopital Tenon /ID# 239179, Paris
  - Institut Gustave Roussy /ID# 267415, Villejuif, Île-de-France Region
- Germany (10):
  - Thoraxklinik Heidelberg gGmbH /ID# 239656, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 238331, Mannheim, Baden-Wurttemberg
  - Asklepios Fachkliniken München-Gauting /ID# 272768, Gauting, Bavaria
  - Universitaetsklinikum Giessen /ID# 252973, Giessen, Hesse
  - Klinikum Kassel /ID# 240142, Kassel, Hesse
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 274719, Dresden, Saxony
  - Universitaetsklinikum Jena /ID# 239661, Jena, Thuringia
  - Charite Universitaetsmedizin Berlin Campus Virchow-Klinikum /ID# 234247, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 239658, Hamburg
  - Haemato-Onkologie Hamburg /ID# 241047, Hamburg
- Greece (5):
  - Henry Dunnant Hospital Center /ID# 267021, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 230824, Athens, Attica
  - Metropolitan Hospital /ID# 232158, Piraeus, Attica
  - Metropolitan Hospital /ID# 239170, Piraeus, Attica
  - Interbalkan Medical Center Of Thessaloniki /ID# 254407, Thessaloniki
- Israel (4):
  - ZIV Medical Center /ID# 238606, Safed, Northern District
  - The Edith Wolfson Medical Center /ID# 233781, Ashkelon, Southern District
  - Soroka University Medical Center /ID# 252711, Beersheba, Southern District
  - Tel Aviv Sourasky Medical Center /ID# 260519, Tel Aviv, Tel Aviv
- Italy (9):
  - Humanitas Istituto Clinico Catanese /ID# 273050, Misterbianco, Catania
  - IRCCS Ospedale San Raffaele /ID# 254376, Milan, Milano
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 252942, Naples, Napoli
  - Azienda Ospedaliera Complesso Ospedaliero San Giovanni-Addolorata /ID# 238618, Rome, Roma
  - I.R.C.C.S Istituto Tumori Giovanni Paolo II /ID# 238696, Bari
  - Azienda Socio Sanitaria Territoriale di Cremona /ID# 238698, Cremona
  - Azienda Ospedaliera Papardo /ID# 258038, Messina
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia /ID# 238473, Perugia
  - ASST Sette Laghi - Ospedale Di Circolo E Fondazione Macchi Varese /ID# 238536, Varese
- Japan (42):
  - NHO Nagoya Medical Center /ID# 246306, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 239990, Nagoya, Aichi-ken
  - Hirosaki University Hospital /ID# 242377, Hirosaki-shi, Aomori
  - National Cancer Center Hospital East /ID# 233775, Kashiwa-shi, Chiba
  - National Hospital Organization Kyushu Medical Center /ID# 238533, Fukuoka, Fukuoka
  - Hospital Of The University Of Occupational And Environmental Health, Japan /ID# 241191, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital /ID# 254900, Kurume-shi, Fukuoka
  - Fukushima Medical University Hospital /ID# 249691, Fukushima, Fukushima
  - Gunma Prefectural Cancer Center /ID# 233723, Ota-shi, Gunma
  - Chugoku Central Hospital /ID# 242970, Fukuyama, Hiroshima
  - Hiroshima University Hospital /ID# 241882, Hiroshima, Hiroshima
  - Hokkaido University Hospital /ID# 241289, Sapporo, Hokkaido
  - Kobe Minimally Invasive Cancer Center /ID# 254131, Kobe, Hyōgo
  - Takarazuka City Hospital /ID# 240786, Takarazuka-shi, Hyōgo
  - NHO Mito Medical Center /ID# 241709, Higashiibaraki-gun, Ibaraki
  - Ibaraki Prefectural Central Hospital /ID# 246145, Kasama-shi, Ibaraki
  - Iwate Medical University Hospital /ID# 239027, Shiwa-gun, Iwate
  - Kitasato University Hospital /ID# 239958, Sagamihara-shi, Kanagawa
  - Yokohama City University Medical Center /ID# 246554, Yokohama, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center /ID# 239052, Yokohama, Kanagawa
  - Kumamoto University Hospital /ID# 241039, Kumamoto, Kumamoto
  - National Hospital Organization Mie Chuo Medical Center /ID# 246659, Tsu, Mie-ken
  - Miyagi Cancer Center /ID# 234198, Natori-shi, Miyagi
  - Sendai Kousei Hospital /ID# 253350, Sendai, Miyagi
  - University of Miyazaki Hospital /ID# 242161, Miyazaki, Miyazaki
  - Nagaoka Red Cross Hospital /ID# 240714, Nagaoka-shi, Niigata
  - Kurashiki Central Hospital /ID# 239344, Kurashiki-shi, Okayama-ken
  - Osaka Habikino Medical Center /ID# 239989, Habikino-shi, Osaka
  - Kansai Medical University Hospital /ID# 233476, Hirakata-shi, Osaka
  - Osaka Metropolitan University Hospital /ID# 238895, Osaka, Osaka
  - Kindai University Hospital /ID# 239085, Sakai-shi, Osaka
  - Fujieda Municipal General Hospital /ID# 255155, Fujieda-shi, Shizuoka
  - Tochigi Cancer Center /ID# 240020, Utsunomiya, Tochigi
  - Juntendo University Hospital /ID# 239932, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital /ID# 251134, Chuo-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center /ID# 246581, Meguro-ku, Tokyo
  - NTT Medical Center Tokyo /ID# 241067, Shinagawa-ku, Tokyo
  - Keio University Hospital /ID# 239506, Shinjuku-ku, Tokyo
  - Toyama University Hospital /ID# 241660, Toyama, Toyama
  - Wakayama Medical University Hospital /ID# 234004, Wakayama, Wakayama
  - Yamagata University Hospital /ID# 240815, Yamagata, Yamagata
  - Yamaguchi - Ube Medical Center /ID# 258779, Ube-shi, Yamaguchi
- Mexico (3):
  - O.P.D. Hospital Civil de Guadalajara /ID# 238488, Guadalajara, Jalisco
  - Centro de Investigacion Clínica Chapultepec SA de CV /ID# 231928, Morelia, Michoacán
  - Clinical Research & Oncology Oaxaca /ID# 231883, Oaxaca City
- Netherlands (4):
  - Ziekenhuis St. Jansdal /ID# 251932, Harderwijk, Gelderland
  - Maastricht Universitair Medisch Centrum /ID# 233932, Maastricht, Limburg
  - Isala /ID# 238846, Zwolle, Overijssel
  - HagaZiekenhuis /ID# 243693, The Hague, South Holland
- Poland (5):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeyla /ID# 262489, Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Bada /ID# 262095, Warsaw, Masovian Voivodeship
  - MRUK-MED I Sp. z o.o. /ID# 239363, Rzeszów, Podkarpackie Voivodeship
  - Warminsko-Mazurskie Centrum Chorob Pluc w Olsztynie /ID# 239025, Olsztyn, Warmian-Masurian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki /ID# 239024, Lodz, Łódź Voivodeship
- Portugal (5):
  - Fundacao Champalimaud /ID# 241925, Lisbon, Lisbon District
  - Centro Hospitalar Universitario do Porto, EPE - Hospital Santo Antonio /ID# 241572, Porto
  - Hospital CUF Porto /ID# 241570, Porto
  - IPO Porto FG, EPE /ID# 241569, Porto
  - Unidade Local de Saude Sao Joao, EPE /ID# 241930, Porto
- Romania (8):
  - Spitalul Pelican /ID# 254066, Oradea, Bihor County
  - Cardiomed Srl /Id# 255320, Cluj-Napoca, Cluj
  - Sc Oncolab Srl /Id# 239105, Craiova, Dolj
  - Institutul Regional de Oncologie /ID# 254065, Iași, Iaşi
  - SC RTC Radiology Therapeutic Center SRL /ID# 240744, Otopeni, Ilfov
  - Oncocenter - Oncologie Clinica Srl /Id# 239103, Timișoara, Timiș County
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL /ID# 240826, Brasov
  - S.C. Sigmedical Services SRL /ID# 239108, Suceava
- Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 230084, Banská Bystrica, Banská Bystrica Region, Slovakia
- South Africa (3):
  - Wits Clinical Research /ID# 230841, Johannesburg, Gauteng
  - Sandton Oncology Medical Group PTY Ltd /ID# 230843, Johannesburg, Gauteng
  - Steve Biko Academic Hospital /ID# 230883, Pretoria, Gauteng
- South Korea (10):
  - National Cancer Center /ID# 260663, Goyang-si, Gyeonggido
  - CHA Bundang Medical Center /ID# 233318, Seongnam, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 256942, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 233319, Suwon, Gyeonggido
  - Gyeongsang National University Hospital /ID# 234244, Jinju, Gyeongsangnam-do
  - Pusan National University Yangsan Hospital /ID# 257836, Yangsan, Gyeongsangnam-do
  - Chungbuk National University Hospital /ID# 257891, Cheongju-si, North Chungcheong
  - Kangbuk Samsung Hospital /ID# 233711, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 256941, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 233710, Seoul, Seoul Teugbyeolsi
- Spain (9):
  - CHU Insular-Materno Infantil /ID# 255094, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Fundacion Alcorcon /ID# 255100, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada /ID# 255093, Fuenlabrada, Madrid
  - Hospital Nuestra Senora de Sonsoles /ID# 255102, Ávila
  - UOMi Cancer Center - Clinica Tres Torres /ID# 240584, Barcelona
  - Hospital Universitario Dexeus - Grupo Quironsalud /ID# 255105, Barcelona
  - Hospital Universitario de Jaen /ID# 240588, Jaén
  - Hospital Universitario 12 de Octubre /ID# 240176, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 240378, Valencia
- Sweden (2):
  - Karolinska University Hospital Solna /ID# 229853, Solna, Stockholm County
  - Sahlgrenska Universitetssjukhuset /ID# 229943, Gothenburg, Västra Götaland County
- Taiwan (8):
  - E-DA Cancer Hospital /ID# 239718, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 238378, Taipei City, Taipei
  - Changhua Christian Hospital /ID# 238394, Changhua City, Changhua County
  - National Taiwan University Hospital - Hsinchu branch /ID# 238393, Hsinchu
  - Hualien Tzu Chi Hospital /ID# 238398, Hualien City
  - Chung Shan Medical University Hospital /ID# 238444, Taichung
  - Mackay Memorial Hospital /ID# 238392, Taipei
  - Taipei Medical University Hospital /ID# 238380, Taipei
- Turkey (Türkiye) (12):
  - Memorial Ankara Hastanesi /ID# 234212, Çankaya, Ankara
  - Izmir Ekonomi Universitesi Ozel Medicalpoint Hastanesi /ID# 234209, Cordaleo, İzmir
  - Adana Sehir Egitim ve Arastirma Hastanesi /ID# 255638, Adana
  - Adana Acıbadem Hospital /ID# 234208, Adana
  - Medical Park Seyhan Hastanesi /ID# 255637, Adana
  - Ankara City Hospital /ID# 234210, Ankara
  - Inonu Universitesi Turgut Ozal /ID# 234038, Battalgazi/malatya
  - Uludag University Medical Faculty /ID# 234205, Bursa
  - Dicle Universitesi Tip /ID# 234036, Diyarbakır
  - Bagcilar Medipol Mega Universite Hastanesi /ID# 234211, Istanbul
  - Ege University Medical Faculty /ID# 234039, Izmir
  - Dr. Suat Seren Gogus Has /ID# 262291, Izmir
- United Kingdom (6):
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 254342, London, Greater London
  - University College London Hospital /ID# 249407, London, Greater London
  - Nottingham City Hospital /ID# 254707, Nottingham, Nottinghamshire
  - University Hospitals Birmingham NHS Foundation Trust /ID# 258141, Birmingham
  - The Royal Marsden NHS Foundation Trust /ID# 246974, London
  - The Christie Hospital /ID# 243422, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/